CLINICAL TRIAL: NCT00569829
Title: A Randomized, Controlled Trial of Modular CBT for Child Anxiety Disorders in Elementary School Settings
Brief Title: Modular Cognitive Behavioral Therapy for the Treatment of Child Anxiety Disorders in Elementary School Settings
Acronym: KATES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey J. Wood, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G04-06-117-04
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Separation Anxiety Disorder; Generalized Anxiety Disorder; Social Phobia
Keywords: cognitive behavioral therapy; anxiety disorders; school-based intervention; randomized, controlled trial
MeSH Terms: conditions — Anxiety, Separation; Generalized Anxiety Disorder; Phobia, Social; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cognitive behavioral therapy
  Interventions: Behavioral: cognitive behavioral therapy
- 2 (No Intervention): Waitlist

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — 1 to 16 weekly sessions of modular cognitive behavioral therapy, each lasting 60-80 minutes
  Arms: 1

SUMMARY:
Although cognitive behavioral therapy (CBT) has been found to be efficacious in the treatment of child anxiety disorders, little progress has been made in the dissemination of such treatments to real-world practice settings. Clinical trials conducted in practice settings can demonstrate the degree to which evidence-based treatments are appropriate for larger scale dissemination. This study evaluates CBT as a treatment for child anxiety disorders in the elementary school clinic setting. A randomized, controlled trial design has been employed, comparing immediate treatment and a three-month waitlist. The trial is being conducted in several Los Angeles area elementary schools and is only available to children in these particular schools. To ensure that the CBT intervention is flexible and capable of matching the characteristics of various school settings, clinicians, and referred children, a modular treatment approach is employed. The study design includes elements to ensure high quality data, such as the use of independent evaluators and tests of treatment fidelity. Children, ages 5 to 12 years, are referred by teachers and staff or are identified as having high anxiety in concurrent studies. All participating children have DSM-IV diagnoses of separation anxiety disorder, generalized anxiety disorder, or social phobia, according to a semi-structured diagnostic interview. Therapy and clinical supervision is provided by the research team. It is hypothesized that children receiving immediate treatment will have significantly lower anxiety scores than children assigned to the waitlist at the posttreatment/postwaitlist assessment. If results are favorable, further exploration of dissemination of CBT into school clinic settings may be indicated.

ELIGIBILITY:
Inclusion Criteria:

* The child meets DSM-IV criteria for separation anxiety disorder (SAD), social phobia, or generalized anxiety disorder (GAD) based on a diagnostic interview
* The child is not taking any psychiatric medication at the initial assessment, or is taking a stable dose of psychiatric medication (i.e., at least one month at a stable dose prior to the baseline assessment)
* If medication is being used, children will maintain that dose throughout the study

Exclusion Criteria:

* The child is currently in psychotherapy
* The family is currently in family therapy or a parenting class
* The child begins taking psychiatric medication or increases his/her dose of medication during the intervention
* For any reason the child or parents appear unable to participate in the intervention program.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2004-01; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Clinician's Global Impressions-Improvement (CGI) scale | Posttreatment / postwaitlist

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule IV: Child and Parent Version | Posttreatment / postwaitlist

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Wood, PhD, Principal Investigator — University of California, Los Angeles